CLINICAL TRIAL: NCT06242483
Title: The ELFIE-HYPERTENSION Randomized Clinical Trial
Brief Title: The ELFIE-HYPERTENSION
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Elfie Pte. Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ELFIE
Record Dates: First submitted 2024-01-29; First posted 2024-02-05 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Hypertension
Keywords: Blood pressure; Digital health intervention
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants will be instructed not to mention their allocated group to the outcome assessor until the end of the follow-up visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care group (No Intervention): Patients randomized to usual care will receive standard care, in which hypertension treatment will be provided according to local practices and will not have access to the Elfie solution. Additionally, they will be requested not to access/use other mobile phone apps or participate in any kind of digital health intervention related to hypertension treatment during the trial.
- Digital health intervention group (Elfie solution) (Experimental): Patients randomized to digital health intervention group will receive standard care plus the Elfie solution. Participants randomized to the Elfie solution will be instructed to download the Elfie app and will receive training on how to register in the app and on how to use all the app features. Participants will be then instructed to use the app according to the monitoring plan created by the app for the following 6 months.
  Interventions: Other: Elfie Solution

INTERVENTIONS:
Other: Elfie Solution — The Elfie solution was designed to improve knowledge, adherence, and the quality of care for patients with cardiovascular diseases. The Elfie solution comprises a mobile phone app with the following features related to hypertension:
  1. Personalized monitoring plan based on health conditions to guide frequency of monitoring of blood pressure, weight, and step count
  2. Digital pillbox with daily medication-taking reminders and refill reminders
  3. Clinical measurements graphs for BP, weight, medical adherence and step count
  4. Newsfeed with short videos and texts related to cardiovascular diseases
  5. Digital coach - Artificial intelligence technology that provides information via a chatbox as well as feedback information via personalized videos. This feature does not provide medical advice.
  6. Connection with a health app or wearable for step count
  7. Possibility of family peer support
  8. Gamification through the Elfie rewards scoring system
  Arms: Digital health intervention group (Elfie solution)

SUMMARY:
The ELFIE-HYPERTENSION randomized clinical trial is an academic-led, collaborative, pragmatic, randomized, open-label, parallel arm, multicenter, trial evaluating whether a digital health intervention based on the Elfie solution compared with usual care will reduce systolic blood pressure in individuals with hypertension.

DETAILED DESCRIPTION:
The ELFIE-HYPERTENSION randomized clinical trial is an academic-led, collaborative, pragmatic, randomized, open-label, parallel arm, multicenter, trial evaluating whether a digital health intervention based on the Elfie solution compared with usual care will reduce systolic blood pressure in individuals with hypertension. The study will also evaluate whether this digital health intervention compared to usual care will improve diastolic blood pressure, adherence to anti-hypertensive medication, anti-hypertensive treatment intensification, body mass index, hypertension knowledge, self-care, quality of life, and the need for unscheduled cardiovascular-related medical assessment.

The hypothesis is that the Elfie solution will improve blood pressure control in individuals with hypertension

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 75 years
* Male and female patients
* Hypertension diagnosis based on the local guidelines criteria
* Uncontrolled blood pressure (systolic blood pressure ≥ 140 mmHg) on the screening visit
* Patients in whom medication adherence needs to be improved according to the healthcare provider clinical judgment
* Use of at least 1 anti-hypertensive medication
* Ownership of an active smartphone with operational system iOS (version 13.0 or later) or Android (version 8.0 or later) with access to the internet on 3G, 4G or 5G
* Ability to use a smartphone app

Exclusion Criteria:

* Refusal to provide written informed consent
* Current use of a health app with the aim to improve medication adherence and blood pressure control
* Illiteracy to read in the local language
* Known cognitive decline, dementia, or diagnosis of severe psychiatric conditions (depression, schizophrenia, bipolar disorder)
* Known use of illicit drugs or alcoholism
* Current participation in a cardiovascular randomized clinical trial
* Life expectancy < 1 year

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 930 (Actual)
Dates: Start 2024-06-14 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Office systolic blood pressure (SBP) | 6-months
  Mean systolic blood pressure in the office

SECONDARY OUTCOMES:
Percentage (%) of participants achieving office SBP < 140mmHg | 6-months
  Percentage (%) of participants achieving office SBP < 140mmHg
Percentage (%) of participants achieving office SBP < 130mmHg | 6-months
  Percentage (%) of participants achieving office SBP < 130mmHg
Office diastolic blood pressure (DBP) | 6-months
  Mean diastolic blood pressure in the office
Percentage (%) participants achieving DBP < 90mmHg | 6-months
  Percentage (%) participants achieving DBP < 90mmHg
Percentage (%) participants achieving DBP < 80mmHg | 6-months
  Percentage (%) participants achieving DBP < 80mmHg
Anti-hypertensive treatment intensification | 6-months
  Intensification of anti-hypertensive treatment
Body mass index | 6-months
  Mean body mass index
Adherence to anti-hypertensive medication measured by the 8-item Morisky Medication | 6-months
  8-item Morisky Medication Adherence Scale (MMAS)
Level of hypertension knowledge measured by the Hypertension Knowledge-level scale | 6-months
  Hypertension Knowledge-level scale (HK-LS)
Level of hypertension-related self-care measured by the Self-care of Hypertension | 6-months
  Self-care of Hypertension Inventory (SC-HI)
Quality of life measured by the SF-12 questionnaire | 6-months
  SF-12 questionnaire
CV-related unscheduled visits to the doctor's office or emergency room | 6-months
  Number of unscheduled visits

OTHER OUTCOMES:
Duration of app use | 6-months
  Mean time between first and last logins in the app during study period
Frequency of app use | 6-months
  Mean number logins in the app
Mean duration (minutes) of login sessions | 6-months
  Mean duration (minutes) of login sessions
% intervention participants who entered at least 1 blood pressure measurement in the app | 6-months
  % intervention participants who entered at least 1 blood pressure measurement in the app
Mean number blood pressure measurements entered in the app | 6-months
  Mean number blood pressure measurements entered in the app
Mean systolic blood pressure entered in the app | 6-months
  Mean systolic blood pressure entered in the app (both manually entered and automatically transmitted via Bluetooth)
Mean diastolic blood pressure entered in the app | 6-months
  Mean diastolic blood pressure entered in the app (both manually entered and automatically transmitted via Bluetooth)
% intervention participants who entered at least 1 medication (any medication) in the app | 6-months
  % intervention participants who entered at least 1 medication (any medication) in the app
% intervention participants who entered at least 1 anti-hypertensive medication in the app | 6-months
  % intervention participants who entered at least 1 anti-hypertensive medication in the app
Mean number medications entered in the app | 6-months
  Mean number medications entered in the app
Types of medications entered in the app | 6-months
  Anti-hypertensive, anti-diabetic, lipid-lowering medications
% adherence to medications in the app | 6-months
  % adherence to medications in the app
% intervention participants who entered at least 1 weight measurement in the app | 6-months
  % intervention participants who entered at least 1 weight measurement in the app
Mean number weight measurements entered in the app | 6-months
  Mean number weight measurements entered in the app
Mean weight entered in the app | 6-months
  Mean weight entered in the app
% intervention participants who connect the Elfie app with a health app for step count | 6-months
  % intervention participants who connect the Elfie app with a health app for step count
Mean number daily steps | 6-months
  Mean number daily steps
% intervention participants who used the digital coach feature at least once | 6-months
  % intervention participants who used the digital coach feature at least once (both the chatbox and the personalized videos)
Mean number of times the digital coach feature was used | 6-months
  Mean number of times the digital coach feature was used (both the chatbox and the personalized videos)
% intervention participants who used the rewards feature | 6-months
  % intervention participants who used the rewards feature
Mean number of times the rewards feature was used | 6-months
  Mean number of times the rewards feature was used
% intervention participants who used the family support feature | 6-months
  % intervention participants who used the family support feature
% intervention participants who used monitoring features for other diseases (diabetes, dyslipidemia, angina) | 6-months
  % intervention participants who used monitoring features for other diseases (diabetes, dyslipidemia, angina)

CONTACTS AND LOCATIONS:
Overall Officials: Karla Santo, MD, Phd, Principal Investigator — karla.santo@einstein.br
Locations (16):
- Brazil (11):
  - Hosp. Universitário UFG, Goiânia, Goiás
  - Hospital Municipal Aparecida de Goiânia, Goiânia, Goiás
  - NF. Pacheco Cardiologia Humanizada, Belém, Pará
  - Rede AME Saúde, Recife, Pernambuco
  - Hospital Universitário Pedro Ernesto, Rio de Janeiro, Rio de Janeiro
  - Clínica do Coração - JMF, Aracaju, Sergipe
  - Hospital Universitário São Francisco na Providência de Deus, Bragança Paulista, São Paulo
  - Centro de Pesquisa Clínica de Guarulhos, Guarulhos, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo, São Paulo
  - CETRUS - Diagnostica LTDA, São Paulo, São Paulo
  - Elizabeth Do Espirito Santo Eireli, Votuporanga, São Paulo
- Vietnam (5):
  - 354 Military Hospital, Hanoi
  - National Geriatric Hospital, Hanoi
  - District 4 Hospital, Ho Chi Minh City
  - Gia Dinh hospital, Ho Chi Minh City
  - Nguyen Tri Phuong Hospital, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: No